CLINICAL TRIAL: NCT03065452
Title: Sagittal Imbalance and Lumbar Stenosis Surgery: Decompression Without Implant
Acronym: CLE/EOS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MADKOURI-BEAURAIN 2016
Record Dates: First submitted 2017-01-27; First posted 2017-02-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lumbar Stenosis, Familial
MeSH Terms: conditions — Lumbar Stenosis, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent open decompression surgery: Observational study on patients who underwent open decompression surgery

SUMMARY:
Lumbar stenosis (LSS) is the most frequent degenerative lumbar disease and is the most frequent indication for spinal surgery. When non-invasive treatments fail, decompression surgery is the gold standard therapy for the majority of patients and generally improves symptoms.

However, few studies have investigated the improvement in posture (radiological parameters) after surgery. In lumbar stenosis, patients may present a forward leaning posture (to relieve pain), which is responsible for sagittal imbalance.

The aim of this prospective study was to evaluate the repercussions of decompression surgery on sagittal balance and to compare these with aux clinical results. investigators included patients operated on for isolated lumbar canal stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms and signs of neurogenic claudication and radiological signs of central lumbar stenosis;
2. Patients undergoing open decompression surgery ≤ 3 levels,
3. All patients with symptoms that did not respond to at least 3 months of non-invasive treatment.

Exclusion Criteria:

Patients were excluded from the study if they had one or several of the following clinical and/or radiological criteria:

1. spondylolisthesis (disc slip > 5 mm),
2. criteria showing instability (variation of > 10° in the angle formed by the vertebral endplates on dynamic images).
3. scoliosis (Cobb angle > 20 °).
4. Patients lost to follow-up were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients who underwent open decompression surgery (laminotomy) were prospectively included in this study
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Vertical sagittal axis | 12 months
  Evaluation of sagittal parameters

SECONDARY OUTCOMES:
radiographic evaluation with EOS | 12 months
  Use of the EOS system and 3D SterEOS software o carry out very precise measurements and 3D reconstructions by bone modeling which give access to new parameters
Functional Interest | 12 months
  Stenosis self-questionnaire (Zurich Claudication Questionnaire)
Sagittal parameters | 12 months
  PI (pelvic incidence) in degrees,
Sagittal parameters | 12 months
  SS (sacral slope) in degrees
Sagittal parameters | 12 months
  PT (pelvic tilt) in degrees
Sagittal parameters | 12 months
  LL (lumbar lordosis) in degrees
Sagittal parameters | 12 months
  TK in degrees
Sagittal parameters | 12 months
  TPA (T1 Pelvic Angle) in degrees
Sagittal parameters | 12 months
  C7 Barrey's ratio as a percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Dijon, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Madkouri R, Brauge D, Vidon-Buthion A, Fahed E, Mourier KL, Beaurain J, Grelat M. Improvement in Sagittal Balance After Decompression Surgery without Fusion in Patients with Degenerative Lumbar Stenosis: Clinical and Radiographic Results at 1 Year. World Neurosurg. 2018 Jun;114:e417-e424. doi: 10.1016/j.wneu.2018.03.002. Epub 2018 Mar 10. PMID 29530708